CLINICAL TRIAL: NCT04593121
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single- and Multiple-Ascending-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB107 in Healthy Adult Participants
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BIIB107 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 271HV101
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1A (Experimental): Participants will receive Dose 1 of BIIB107 or placebo subcutaneous (SC) on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 2A (Experimental): Participants will receive Dose 2 of BIIB107 or placebo SC on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 3A (Experimental): Participants will receive Dose 3 of BIIB107 or placebo SC on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 4A (Experimental): Participants will receive Dose 4 of BIIB107 or placebo SC on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 7A (Experimental): Participants will receive Dose 5 of BIIB107 or placebo SC on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 5A (Experimental): Participants will receive Dose 5 of BIIB107 or placebo intravenous (IV) on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 8A (Experimental): Participants will receive Dose 6 of BIIB107 or placebo SC on Day 1.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 1B (Experimental): Participants will receive multiple doses of BIIB107 or placebo SC on approximately 4 dosing days.
  Interventions: Drug: BIIB107; Drug: Placebo
- Cohort 2B (Experimental): Participants will receive multiple doses of BIIB107 or placebo SC on approximately 4 dosing days.
  Interventions: Drug: BIIB107; Drug: Placebo

INTERVENTIONS:
Drug: BIIB107 — Administered as specified in the treatment arm.
Drug: Placebo — Administered as specified in the treatment arm.

SUMMARY:
The primary objective is to determine the safety and tolerability of single and multiple ascending subcutaneous (SC) doses and a single intravenous (IV) dose of BIIB107 in healthy adult participants. The secondary objectives are to characterize the single-dose pharmacokinetic (PK) of SC and IV BIIB107 in healthy adult participants and to characterize the multiple-dose PK of SC BIIB107 in healthy adult participants.

DETAILED DESCRIPTION:
BIIB107 is a monoclonal antibody (mAb) that targets alpha-4 integrins and is currently in development for people with multiple sclerosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2), inclusive, and must weigh at least 55 kilogram (kg)
* All women of childbearing potential must practice highly effective contraception during the study and for a period of 90 days, which is expected to be more than 5 half-lives of BIIB107. Men must practice effective contraception during the study and for a period of 5 half-lives of BIIB107 or 90 days after their last dose of study treatment. In addition, participants should not donate sperm or eggs during the study and for at least 5 half-lives of BIIB107 or 90 days after their last dose of study treatment
* Negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction test at Screening and Check-in/admission.

Key Exclusion Criteria:

* History of or positive test result at Screening for human immunodeficiency virus (HIV-1/HIV-2) antibodies
* Positive test result at Screening for hepatitis C virus (HCV) antibody (Ab).
* Current hepatitis B infection (defined as per protocol) and participants with immunity to hepatitis B from previous natural infection (defined as negative hepatitis B surface antigen [HBsAg], positive hepatitis B surface antibody [HBsAb], and positive total hepatitis B core antibody [HBcAb]).
* Signs of active herpes simplex type 1 and 2 or varicella within 4 weeks prior to randomization
* Evidence of current SARS-CoV-2 infection within 4 weeks prior to Screening, at Screening, between Screening and inpatient admission (Day -1), or at admission (Day -1), including but not limited to a fever (temperature >37.5°C), new and persistent cough, breathlessness, or loss of taste or smell, per the judgement of the Investigator.
* Close contact with an individual with coronavirus disease 2019 (COVID-19) infection within 14 days prior to admission (Day -1). Close contact is defined as being within 6 feet of an infected person as confirmed via laboratory assessment for at least 15 minutes within 2 days of symptom onset (or within 2 days of specimen collection for COVID-19 testing for close contact with asymptomatic person).
* History of tuberculosis (TB) or positive QuantiFERON® TB Gold test or, if the QuantiFERON TB Gold test is not available, a positive purified protein derivative (PPD/Mantoux test; positive PPD/Mantoux test is defined as ≥5 millimeter (mm) of induration [size of raised lump, not redness])
* John Cunningham virus (JCV) seropositivity at Screening (for potential participants enrolling in Part B)
* Ongoing or past malignancy, carcinoma in situ, or high-grade dysplasia (with the exception of no more than 1 basal cell carcinoma or squamous cell carcinoma that was completely excised and cured at least 12 months prior to randomization)
* History of severe allergic or anaphylactic reactions or history of allergic reactions that, in the opinion of the Investigator, is likely to be exacerbated by any component of the study treatment.
* Any prior exposure to mAbs, Fc-fusion proteins, or the following immunomodulator therapies per investigator judgement: natalizumab or any other anti-α4 integrin antibodies, anti-CD20, sphingosine-1-phosphate receptor modulators, or fumarate therapies.
* Any previous exposure to immunosuppressants (in particular mitoxantrone, methotrexate, azathioprine, cyclophosphamide, and mycophenolate mofetil). Any corticosteroid use should be discussed with the Sponsor prior to enrollment
* Part B only: Women of childbearing potential.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs): Single Ascending Dose (SAD) | Day -1 up to Day 84
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs): Multiple Ascending Dose (MAD) | Day -1 up to Day 169
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUCinf): SAD | Day 1 pre-dose and multiple time-points up to Day 84
Maximum Observed Concentration (Cmax): SAD | Day 1 pre-dose and multiple time-points up to Day 84
Time to Reach Maximum Observed Concentration (Tmax): SAD | Day 1 pre-dose and multiple time-points up to Day 84
Terminal Half-Life (t1/2): SAD | Day 1 pre-dose and multiple time-points up to Day 84
Clearance (CL) for IV Doses: SAD | Day 1 pre-dose and multiple time-points up to Day 84
Apparent Clearance (CL/F) of SC Doses: SAD | Day 1 pre-dose and multiple time-points up to Day 84
Volume of Distribution at Steady State (Vss) for IV Doses: SAD | Day 1 pre-dose and multiple time-points up to Day 84
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) for SC Doses: SAD | Day 1 pre-dose and multiple time-points up to Day 84
Bioavailability (F) of SC Doses: SAD | Day 1 pre-dose and multiple time-points up to Day 84
Absorption Rate Profile of SC Doses: SAD | Day 1 pre-dose and multiple time-points up to Day 84
Maximum Observed Concentration (Cmax): MAD | Day 1 pre-dose and multiple time-points up to Day 169
Time to Reach Maximum Observed Concentration (Tmax): MAD | Day 1 pre-dose and multiple time-points up to Day 169
Area Under the Concentration-Time Curve Over the Dosing Interval (AUCtau): MAD | Day 1 pre-dose and multiple time-points up to Day 169
Trough Concentration (Ctrough): MAD | Day 1 pre-dose and multiple time-points up to Day 169
Terminal Half-Life (t1/2): MAD | Day 1 pre-dose and multiple time-points up to Day 169
Accumulation Ratio (R): MAD | Day 1 pre-dose and multiple time-points up to Day 169
Apparent Clearance (CL/F) of SC Doses: MAD | Day 1 pre-dose and multiple time-points up to Day 169
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) for SC Doses: MAD | Day 1 pre-dose and multiple time-points up to Day 169

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - CenExel Anaheim Clinical Trials, Anaheim, California
  - QPS MRA (Miami Research Associates), Miami, Florida
  - Altasciences Clinical Research, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/